CLINICAL TRIAL: NCT04255238
Title: A Multicenter, Randomized, Double-blind, Double-dummy, Active-controlled, Parallel Group, Phase 3 Trial to Evaluate the Efficacy and Safety of Dual add-on Therapy With Gemigliptin 50 mg and Dapagliflozin 10 mg Added to Metformin Compared to add-on Therapy With Gemigliptin 50 mg in Combination With Metformin or Dapagliflozin 10 mg in Combination With Metformin in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Metformin Alone
Brief Title: A Study to Evaluate the Efficacy and Safety of Dual add-on Therapy With Gemigliptin 50 mg and Dapagliflozin 10 mg Added to Metformin Who Have Inadequate Glycemic Control on Metformin Alone
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LG-GLCL001
Record Dates: First submitted 2020-02-02; First posted 2020-02-05 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LC15-0444; dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gemigliptin 50 mg and Dapagliflozin 10 mg (Experimental): * Subject shoud took 1 tablet of Gemigliptin 50 mg and 1 tablet of Dapagliflozin 10 mg per day
  * Background therapy should be administered keeping the same dosage administered before the study, according to the following criteria: Metformin ≥ 1,000 mg / day
  Interventions: Drug: Gemigliptin 50mg; Drug: Dapagliflozin 10mg
- Gemigliptin 50 mg and Dapagliflozin placebo (Active Comparator): * Subject shoud took 1 tablet of Gemigliptin 50 mg and 1 tablet of Dapagliflozin placebo per day
  * Background therapy should be administered keeping the same dosage administered before the study, according to the following criteria: Metformin ≥ 1,000 mg / day
  Interventions: Drug: Gemigliptin 50mg
- Gemigliptin placebo and Dapagliflozin 10mg (Active Comparator): * Subject shoud took 1 tablet of Gemigliptin placebo and 1 tablet of Dapagliflozin 10 mg per day
  * Background therapy should be administered keeping the same dosage administered before the study, according to the following criteria: Metformin ≥ 1,000 mg / day
  Interventions: Drug: Dapagliflozin 10mg

INTERVENTIONS:
Drug: Gemigliptin 50mg — The subjects should visit a study site 6-7 times during the treatment period for about 24 weeks in total. - Background therapy should be administered keeping the same dosage administered before the study, according to the following criteria: Metformin ≥ 1,000 mg / day
  Other Names: Zemiglo tab 50mg
  Arms: Gemigliptin 50 mg and Dapagliflozin 10 mg; Gemigliptin 50 mg and Dapagliflozin placebo
Drug: Dapagliflozin 10mg — The subjects should visit a study site 6-7 times during the treatment period for about 24 weeks in total. - Background therapy should be administered keeping the same dosage administered before the study, according to the following criteria: Metformin ≥ 1,000 mg / day
  Other Names: Forxiga tab 10mg
  Arms: Gemigliptin 50 mg and Dapagliflozin 10 mg; Gemigliptin placebo and Dapagliflozin 10mg

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of dual add-on therapy with Gemigliptin 50 mg and Dapagliflozin 10 mg added to Metformin compared to add-on therapy with Gemigliptin 50 mg in combination with Metformin or Dapagliflozin 10 mg in combination with Metformin in patients with type 2 diabetes mellitus who have inadequate glycemic control on metformin alone

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus
* Patients upper 19 years old
* Patients who had taken Metformin(≥1000mg/day) more than 8 weeks and who have inadequate blood glucose control
* Patients who have signed an informed consent themselves after receiving explanation about the clinical study
* Patients who are applicable to one of the three in the following.

  1. Surgically infertile patients
  2. Postmenopausal female patients of ≥45 years of age for whom ≥2 years elapsed since their last menstruation
  3. Premenopausal fertile female patients or surgically non-infertile male patients who have agreed to use at least 2 kinds of contraceptive measures (certainly including one of the barrier methods) to avoid pregnancy until 14 days after the last dose of the investigational product

Exclusion Criteria:

* Patients with type 1 diabetes mellitus, Diabetic ketoacidosis, Metabolic acidosis Diabetic coma, Diabetic pre-coma
* Patients with Gestational diabetes, or secondary diabetes
* Patients with NYHA Class II~IV congestive heart failure or arrhythmia requiring treatment
* Patients whose TSH level is out of the normal range and who have thyroidal dysfunction requiring drug therapy
* Patients with positive Serologic results of HBsAg, HCV Ab, HIV Ab test within 4 weeks prior to Visit 1 (Screening) or at Visit 1 (Screening)
* Patients with Body Mass Index(BMI) #40 kg/m2
* Patients who are receiving intravenous iodine contrast agents within 48 hours prior to Visit 1(Screening) or planned during the clinical trial period (eg, intravenous urography, venous cholangiography, angiography, computed tomography using contrast media, etc.).
* Patients with pulmonary embolism, severe pulmonary dysfunction, or who are susceptible to be accompanied by hypoxemia at the time of Visit 1(Screening)
* Patients on clinically significant dehydration, diarrhea, and vomiting at the time of Visit 1(Screening)
* Patients with pituitary insufficiency or adrenal insufficiency at the time of Visit 1(Screening)
* Patients with a history of alcoholism or drug addiction within 1 years prior to Visit 1(Screening)
* Patients with a history of malignant tumors within 5 years prior to Visit 1(Screening). However, patients with basal cell or squamous cell skin cancer, or in situ cervical cancer treated properly can participate in the study.
* Patients with the outcomes of the laboratory tests performed at Visit

  1(Screening) applicable to the criteria below
  * Bilirubin >2 × upper limit of normal(ULN)
  * AST/ALT >3 × ULN
* Patients with a history of hypersensitivity reactions to the drugs below

  * Dipeptidyl-peptidase4(DPP4) inhibitors
  * Sodium/glucose co transport-2(SGLT-2) inhibitor
  * Biguanides
* Patients who were administered the drugs below
* Patients who had been administered anti-obesity drugs within 12 weeks prior to Visit 1(Screening)
* Patients who have undergone bariatric surgery within the 1 year prior to Visit 1 (Screening) or are scheduled during the trial
* Patients with a genetic problems such as Galactose intolerance, Lapp lactose deficiency, Glucose-galactose malabsorption)
* Female patients who are pregnant or lactating
* Patients who have an experience of participation in another clinical study within 12 weeks prior to Visit1(screening)
* Patients who are otherwise considered to be ineligible for this study on investigators' judgment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Estimated)
Dates: Start 2020-06-30 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Chages from baseline HbA1c at Week24 | Baseline to Week24

IPD SHARING:
Plan to Share IPD: No